CLINICAL TRIAL: NCT01843764
Title: Efficacy of Plasmodium Falciparum Specific Rapid Diagnostic Tests for Assessment of Initial Clearance and Detection of Recurrent Infections After Antimalarial Treatment
Brief Title: Rapid Diagnostic Tests for Assessment of Initial Clearance and Detection of Recurrent Malaria Infections
Status: Completed | Type: Observational
Sponsor: Anders Björkman (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Sponsor-Investigator, Anders Björkman, Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Other Study IDs: RDT-ClearTZ1; KI-MUHAS1 (Registry Identifier: RDT-ClearTZ1)
Record Dates: First submitted 2013-02-15; First posted 2013-05-01 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: RDT; malaria; treatment follow up; diagnosis
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole capillary blood collected for Rapid Diagnostic tests, microscopy and PCR
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- children with malaria: Tanzanian children between 6-59 months with an uncomplicated P.falciparum monoinfection, followed after arthemeter-lumefantrine treatment according to national treatment guidelines
  Interventions: Device: HRP2 and LDH based rapid diagnostic tests for P.falciparum

INTERVENTIONS:
Device: HRP2 and LDH based rapid diagnostic tests for P.falciparum
  Other Names: ParaHit (HRP2); CareStart (pLDH)

SUMMARY:
The aim of the study was to follow clearance of malaria infections and detection of new malaria episodes after initiation of antimalarial treatment in Tanzanian children. For this purpose the investigators used five diagnostic tools, 2 Rapid Diagnostic tests based on Histidine Rich Protein 2(HRP2) and Lactate dehydrogenase(LDH), 2 microscopical methods and one polymerase chain reaction (PCR). The investigators followed the 53 enrolled children during 42 days.

ELIGIBILITY:
Inclusion Criteria:

* children between 6-59 months
* fever (≤37.5 C) or history of fever during the preceding 24 hours
* confirmed P.falciparum monoinfection
* uncomplicated malaria
* parasite density between 2000-250.000/µL
* willing/able to comply with the 42 day follow up
* informed concent from patient/guardian

Exclusion Criteria:

* children with history of antimalaria drug intake within the last two weeks
* symptoms / signs of severe disease

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with fever visiting primary health care units in malaria endemic area
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Clearance time with five diagnostic tests | 2009 June to 2012 May (up to day 42)
  Children were followed up on 9 occasions until day 42. Mean and median time until clearance after initiation of arthemeter-lumefantrine treatment was measured for HRP2 based Rapid diagnostic tests, LDH-based Rapid diagnostic tests, Giemsa and Acridine Orange stained microscopy and real-time PCR.
Detection of recurrent infection with HRP2 and LDH-based Rapid diagnostic tests during follow up | 2009 June to 2012 May (up to day 42)
  Ability to detect recurrent malaria infection with the HRP2 and LDH-Rapid diagnostic tests during the 42 days of follow up was studied through comparing them with three other diagnostic tests.

SECONDARY OUTCOMES:
Efficiency of P.falciparum specific rapid diagnostic tests | 2009 June to 2012 May (up to day 42)
  Efficiency of two rapid diagnostic tests based on two different antigens for diagnosis and treatment follow up among children <5 years in a moderately high endemic area was determined. Specificity and false positivity rate for HRP2 and LDH based rapid diagnostic tests are calculated against Giemsa stained microscopy and PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Björkman, Professor, Study Director — Karolinska Institutet
Locations (2):
- Tanzania (2):
  - Mlandizi Health Centre and Fukayosi dispencary, Dar es Salaam, Kibaha and Bagamoyo District
  - Muhimbili University of Health Allied Science, Dar es Salaam

REFERENCES:
- [Derived] Aydin-Schmidt B, Mubi M, Morris U, Petzold M, Ngasala BE, Premji Z, Bjorkman A, Martensson A. Usefulness of Plasmodium falciparum-specific rapid diagnostic tests for assessment of parasite clearance and detection of recurrent infections after artemisinin-based combination therapy. Malar J. 2013 Oct 1;12:349. doi: 10.1186/1475-2875-12-349. PMID 24079306